CLINICAL TRIAL: NCT01552824
Title: Randomized Controlled Trial of Fetal Cystoscopy Versus Vesico-amniotic Shunting in Severe Lower Urinary Tract Obstructions
Brief Title: Fetal Cystoscopy Versus Vesico-amniotic Shunting in Severe Lower Urinary Tract Obstructions
Acronym: CYSTUO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rodrigo Ruano, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0853/11; 0853/11 (Other: CAPPesq)
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Lower Urinary Tract Obstructive Syndrome
Keywords: LUTO; posterior urethral valves; urethral atresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vesico-amniotic shunt (Experimental): In this arm, patients will be randomly selected to undergo vesico-amniotic shunting.
  Interventions: Procedure: Vesico-amniotic shunt
- CYSTO (Experimental): In this arm, all patients will be randomly selected for fetal cystoscopy.
  Interventions: Procedure: CYSTO

INTERVENTIONS:
Procedure: CYSTO — Fetal cystoscopy will be performed by introducing a 2.2mm sheath with 1.0mm fetoscope into fetal bladder under ultrasound guidance. The fetoscope will be advanced and the posterior urethral valves will be coagulated by ND:YAG laser. If urethra atresia was diagnosed, a vesico-amniotic shunting will be placed. Maternal anesthesia will be conducted by epidural anesthesia and fetal anesthesia will be conducted by injecting fentanyl (15 μg/Kg) and pancuronium (2 mg/Kg) under ultrasound guidance of a 22 gauge needle into fetal arm muscle.
  Arms: CYSTO
Procedure: Vesico-amniotic shunt — In this arm, all patients randomly selected for this treatment will undergo vesico-amniotic shunting under ultrasound guidance. Maternal anesthesia will be conducted by epidural anesthesia and fetal anesthesia will be conducted by injecting fentanyl (15 μg/Kg) and pancuronium (2 mg/Kg) under ultrasound guidance of a 22 gauge needle into fetal arm muscle.
  Arms: Vesico-amniotic shunt

SUMMARY:
There are two options of fetal treatment in cases of severe lower urinary tract obstructions: the vesico-amniotic shunting and fetal cystoscopy. There is no study confirming the effectiveness of these treatment, specially comparing both techniques. The present study aims to investigate the effectiveness of these treatments.

DETAILED DESCRIPTION:
Objectives: To evaluate the effectiveness of fetal cystoscopy for the diagnosis and therapy of the posterior urethral valves and to compare with the results of vesicoamniotic shunting.

Outcomes: Accuracy of the prenatal cystoscopic diagnosis of posterior urethral valves, neonatal and infant survival (6 and 12 months), as well as normal renal function during the same ages.

Study design: Randomized controlled trial. Methods: Pregnant women whose fetuses have isolated and severe lower urinary tract obstruction (LUTO) with (oligohydramnios and severe hydronephrosis) will be invited to participate in the present study. Patients will be randomized into the fetal cystoscopic group (CYSTO) vs vesico-amniotic shunting (VAS). The investigators intend to enroll 30 patients in each group (a total of 60). All patients will be followed by fetal ultrasound each 15 days. Besides, these infants will be followed up to one year of age. Maternal and obstetrical complications are going to be evaluated as well as neonatal and infant survival and the renal function.

ELIGIBILITY:
Inclusion Criteria:

* single pregnancy
* male fetuses
* gestational age dating by ultrasound examination performed before 20 weeks
* confirmed severe LUTO (see details before)
* severe oligohydramnios (AFI<5.0cm)
* no other structural anomalies by complete fetal anatomy ultrasound scan and fetal echocardiogram
* no abnormal karyotype
* 'favorable' urine analysis (urinary sodium <100 mEq/L, chloride <90 mEq/L, osmolarity <200 mOsm/L) when gestational age >20 weeks

Exclusion Criteria:

* presence of other anomalies diagnosed after fetal intervention
* maternal refusal to participate in the present protocol

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Perinatal survival rate | from fetal period to neonatal perid (up to 28 days after birth)
  The primary outcome is survival from the treatment to the neonatal period (up to 28 days of life). Therefore, the objective is to evaluate the safety and effectiveness of both therapeutic options.
Neonatal renal function | up to 28 days of life
  Renal function will be evaluated by serum creatine and urinalysis in the neonates, as well as by micturating cystourethrography and postnatal cystoscopy after birth up to 28 days of life.

SECONDARY OUTCOMES:
Survival rate at 6 months | Up to 6 months of life
  The survival rate up to 6 months of life will be evaluated.
Renal function at 6 months of life | 6 months of life
  Renal function will be evaluated by serum creatinine, need for dialysis and/or renal transplantation.
Survival rate at 1 year of age | 1 year of age
  The survival rate will be evaluated at 1 year of age.
Renal function at 1 year of age | 1 year of age
  Renal function will be evaluated by serum creatinine, need for dialysis and/or renal transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruano, MD, PhD, Principal Investigator — Faculdade de Medicina da Universidade de Sao Paulo
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Ruano R, Pimenta EJ, Duarte S, Zugaib M. Four-dimensional ultrasonographic imaging of fetal lower urinary tract obstruction and guidance of percutaneous cystoscopy. Ultrasound Obstet Gynecol. 2009 Feb;33(2):250-2. doi: 10.1002/uog.6292. No abstract available. PMID 19173237
- [Background] Ruano R, Duarte S, Bunduki V, Giron AM, Srougi M, Zugaib M. Fetal cystoscopy for severe lower urinary tract obstruction--initial experience of a single center. Prenat Diagn. 2010 Jan;30(1):30-9. doi: 10.1002/pd.2418. PMID 19967749
- [Background] Ruano R, Yoshisaki CT, Salustiano EM, Giron AM, Srougi M, Zugaib M. Early fetal cystoscopy for first-trimester severe megacystis. Ultrasound Obstet Gynecol. 2011 Jun;37(6):696-701. doi: 10.1002/uog.8963. PMID 21337440
- [Background] Morris RK, Ruano R, Kilby MD. Effectiveness of fetal cystoscopy as a diagnostic and therapeutic intervention for lower urinary tract obstruction: a systematic review. Ultrasound Obstet Gynecol. 2011 Jun;37(6):629-37. doi: 10.1002/uog.8981. Epub 2011 May 16. PMID 21374748
- [Background] Ruano R. Fetal surgery for severe lower urinary tract obstruction. Prenat Diagn. 2011 Jul;31(7):667-74. doi: 10.1002/pd.2736. Epub 2011 Mar 17. PMID 21413041